CLINICAL TRIAL: NCT03177044
Title: Behavioural Treatment for Functional Bowel Symptoms in Inflammatory Bowel Disease
Acronym: LIBERATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Vincent's Hospital Melbourne (Other)
Responsible Party: Principal Investigator, Angela Khera, Principal Investigator, St Vincent's Hospital Melbourne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREC/17/SVHM/92
Record Dates: First submitted 2017-06-01; First posted 2017-06-06 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Inflammatory Bowel Diseases; Functional Gastrointestinal Disorders
Keywords: Inflammatory bowel disease, pelvic floor exercise
MeSH Terms: conditions — Inflammatory Bowel Diseases; Gastrointestinal Diseases

STUDY DESIGN:
Intervention Model Description: Prospective cohort
Masking Description: All assessments are conducted by an assessor not providing the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioural treatment (Experimental): 2 to 6 sessions of bowel behavioural training with a pelvic floor physiotherapist
  Interventions: Behavioral: Behavioural treatment

INTERVENTIONS:
Behavioral: Behavioural treatment — 2 to 6 sessions of behavioural training with a pelvic floor physiotherapist
  Other Names: Behavioural training programme

SUMMARY:
The primary aim of the project is to investigate whether a behavioural training programme improves troublesome bowel symptoms, that people with inflammatory bowel disease continue to have, despite their disease being controlled by medication. The other aim is to determine if there are factors which influence how well the training programme works.

People attending an Inflammatory Bowel Disease clinic in a tertiary hospital, with bothersome bowel symptoms despite disease control, will be asked to join the study. This involves 2 to 6 sessions with a pelvic floor trained physiotherapist over a period of 6 months with further follow up at 12 months..

DETAILED DESCRIPTION:
Inflammatory bowel diseases, chiefly Crohn's disease and ulcerative colitis, are chronic gastrointestinal (gut) conditions which tend to flare up some times and be quiet for other periods of time. They are usually controlled by medication. Inflammatory bowel disease is becoming more common, is usually diagnosed at a young age and is lifelong.

A significant number of people with inflammatory bowel disease can have bowel symptoms which are bothersome even when the disease is quiescent. These symptoms include bowel urgency, frequent toileting, incontinence (leakage), constipation (infrequent bowel actions and/or difficulty emptying the bowel), abdominal pain, rectal pain or abdominal bloating. The symptoms can be very embarrassing or stressful, limiting activities and making life less enjoyable.

People with these bowel symptoms, but without inflammatory bowel disease, respond to a type of therapy called behavioural treatment. We don't know yet if this treatment helps people with inflammatory bowel disease.

Behavioural treatment involves learning about how the bowel works, better ways to manage bowel problems and specific exercises to improve bowel control. Specially trained pelvic floor physiotherapists provide 2-6 sessions, over 6 months, of behavioural treatment which may include the use of biofeedback techniques.

Participants will be asked to complete surveys at the beginning and end of treatment and 12 months later.

There are no recognised risks or unwanted side effects caused by behavioural treatment. The benefits are that people with inflammatory bowel disease will have an alternative low cost, low risk treatment which enables them to self-manage bowel symptoms and improve the quality of their life long term.

ELIGIBILITY:
Inclusion Criteria:

* Proven history of inflammatory bowel disease
* Clinical evidence of mild, stable disease or remission
* Mayo score ≤ 4, Harvey Bradshaw index ≤ 7
* Bothersome lower bowel symptoms of any of the following: frequency, urgency, incontinence, difficult evacuation, constipation

Exclusion Criteria:

* Significant medical or psychiatric comorbidity that in the opinion of the investigators would interfere with bowel function or adherence to the protocol
* Clinically significant narcotic or substance abuse that in the opinion of the investigators would interfere with bowel function or adherence to the protocol
* Recognised eating disorder
* Non- English speaking or illiterate
* Pregnancy
* Previous pelvic floor physiotherapy
* Current participant in another trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Patient rating of improvement in symptoms | At study completion, up to 12 weeks
  Proportion of patients achieving a rating of 'moderately improved' or 'substantially improved' on a 7 point Likert scale ranging from 'substantially worse' to 'substantially improved'

SECONDARY OUTCOMES:
Change in Personal assessment of Constipation Symptoms (PAC-SYM) score | From baseline to study completion (up to 12 weeks) and at 1 year
  12 constipation symptoms each rated on a 5 point Likert scale (0=symptom absent to 4 = very severe.
Change in St Marks Faecal Incontinence Score | From baseline to study completion (up to 12 weeks) and at 1 year
  Faecal incontinence symptom score ranging from 0-24
Change in Inflammatory Bowel disease questionnaire (IBDQ) score | From baseline to study completion (up to 12 weeks) and at 1 year
  Disease specific quality of life instrument with 32 questions covering 4 domains - bowel symptoms, systemic symptoms, emotional function, social function
Change in Short Form -36 (SF-36) score | From baseline to study completion (up to 12 weeks) and at 1 year
  Generic quality of life score
Change in Hospital Anxiety and Depression Score (HADS) | From baseline to study completion (up to 12 weeks) and at 1 year
  14 item questionnaire indicating presence of anxiety or depression
Change in Brief Illness Perception Questionnaire score | From baseline to study completion (up to 12 weeks) and at 1 year
  9 item questionnaire designed to assess cognitive and emotional perception of illness
Change in Brief Cope score | From baseline to study completion (up to 12 weeks) and at 1 year
  28 item questionnaire assessing patients' strategies for coping with stress
Change in Inflammatory Bowel Disease Self-efficacy scale (IBD-SES) | From baseline to study completion (up to 12 weeks) and at 1 year
  Disease specific scale with 29 items assessing how well patients believe they are managing their disease
Change in Euro-Qol (EQ-5D) | From baseline to study completion (up to 12 weeks) and at 1 year
  Generic quality of life tool to calculate quality adjusted life years (QALYs)

OTHER OUTCOMES:
Change in Mayo Score | From baseline to study completion (up to 12 weeks) and at 1 year
  Disease activity index for ulcerative colitis
Change in Harvey Bradshaw Index | From baseline to study completion (up to 12 weeks) and at 1 year
  Disease activity index for Crohn's disease
Patient rating of satisfaction | At study completion , up to 12 weeks
  7 point Likert scale rating satisfaction
Change in pelvic floor muscle function | From baseline to study completion (up to 12 weeks)
  Measurement of pelvic floor muscle movement using transperineal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Kamm, MBBS PhD, Study Director — St Vincent's Hospital Melbourne
Locations (1):
- St Vincent's Hospital, Fitzroy, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No